CLINICAL TRIAL: NCT04802174
Title: A Phase I/II Trial of Lurbinectedin With Berzosertib, an ATR Kinase Inhibitor in Small Cell Cancers and High Grade Neuroendocrine Cancers
Brief Title: Lurbinectedin With Berzosertib, an ATR Kinase Inhibitor in Small Cell Cancers and High-Grade Neuroendocrine Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000176; 000176-C
Record Dates: First submitted 2021-03-16; First posted 2021-03-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12-08

CONDITIONS: SCLC; Small Cell Cancer; Advanced Solid Tumor; High Grade Neuroendocrine Cancers
Keywords: SCLC; HGNC; M6620
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — PM 01183; berzosertib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/ Phase I (Experimental): Dose escalation of Berzosertib + lurbinectedin
  Interventions: Drug: Lurbinectedin; Drug: Berzosertib
- 2/ Phase II (Experimental): Berzosertib + lurbinectedin at MTD
  Interventions: Drug: Lurbinectedin; Drug: Berzosertib

INTERVENTIONS:
Drug: Lurbinectedin — Participants meeting inclusion and exclusion criteria will receive lurbinectedin (on day 1) and berzosertib (on day 1 and 2) administered every 21 days (1 cycle), either in the in-patient or out-patient setting, until disease progression or development of intolerable side effects.
Drug: Berzosertib — Participants meeting inclusion and exclusion criteria will receive lurbinectedin (on day 1) and berzosertib (on day 1 and 2) administered every 21 days (1 cycle), either in the in-patient or out-patient setting, until disease progression or development of intolerable side effects.

SUMMARY:
Background:

Small cell lung cancer (SCLC) and high-grade neuroendocrine cancers (HGNEC) are aggressive neuroendocrine cancers. At first, SCLC and HGNEC respond to chemotherapy. But then they relapse quickly and become resistant to treatment. Researchers want to see if a combination of drugs can help.

Objective:

To see if the combination of lurbinectedin and berzosertib may be effective to shrink SCLC and HGNEC tumors, and to find the best dose of the combination.

Eligibility:

Adults ages 18 and older with a solid tumor, SCLC, or HGNEC.

Design:

Participants will get lurbinectedin by intravenous (IV) catheter on Day 1 of each cycle (1 cycle = 21 days). They will get berzosertib by IV on Days 1 and 2 of each cycle.

Participants will continue to receive treatment as long as they are benefiting from treatment.

Participants will have physical exams and blood tests. Their symptoms, medicines, and ability to perform their normal activities will be reviewed.

Participants will have electrocardiograms to test heart function. Sticky pads will be placed on their chest, arms, and legs.

Participants will give blood and hair samples for research. They may have optional tumor biopsies.

Participants will have computed tomography (CT) scans to see if the treatment is effective.

Participants will have a follow-up visit 1 month after treatment ends. Then they will be followed by email or phone for the rest of their life.

DETAILED DESCRIPTION:
Background:

Small cell lung cancer (SCLC) and high-grade neuroendocrine cancers (HGNEC) are aggressive neuroendocrine cancers with poor prognosis. Although responsive to chemotherapy initially, both tumor types relapse quickly and become refractory to treatment within a few months.

Replication stress is an SCLC hallmark, driven by oncogenes that drive rapid and unscheduled proliferation (TP53 and RB1 inactivation, MYC amplification, etc.). HGNECs share similarities in morphology, biologic behavior with SCLC. Treatment paradigms have largely paralleled those established for SCLC.

ATR is the master regulator of replication stress response. Upon activation, the ATR CHK1 signaling leads to cell cycle arrest and promotes replication fork stabilization and restart.

ATR inhibition generates replication stress and disables cell cycle checkpoints to ultimately cause mitotic catastrophe and cell death. Many genotoxic agents currently used in cancer therapy are also potent inducers of replication stress.

Berzosertib is a potent and selective kinase inhibitor of ATR, with demonstrated safety and anti-tumor activity as monotherapy and combination with multiple chemotherapeutics (including platinum, gemcitabine, and topoisomerase inhibitors) in high replication stress tumors.

Lurbinectedin is a recently approved second-line SCLC treatment which forms DNA adducts by covalently binding to the minor groove of DNA that kills cancer cells by inhibiting Pol-II and causing DNA damage

We hypothesize that a combination of ATR kinase inhibition with lurbinectedin will provide an attractive synergistic therapeutic option for SCLC and HGNEC.

Primary objectives:

Phase I: To identify the maximum tolerated dose (MTD) of lurbinectedin in combination with berzosertib.

Phase II: To assess the efficacy with respect to clinical response rate of a combination of lurbinectedin and berzosertib in previously treated participants with SCLC and HGNECs.

Eligibility:

All phases: Participants must be greater than or equal to 18 years of age and have a performance status (ECOG) less than or equal to 2. Participants must not have received chemotherapy or undergone major surgery within 2 weeks and radiotherapy within 24 hours prior to enrollment.

Phase I: Participants with histologically confirmed solid tumors and progression on standard therapies. Participants with evaluable, but not measurable disease will be eligible for Phase I.

Phase II: Participants with histological confirmation of SCLC or HGNEC. Participants must have measurable disease to be eligible for Phase II.

Design:

This is a Phase I/II, open label clinical trial identifying the maximum tolerated dose (MTD) of lurbinectedin in combination with berzosertib in a phase I trial, and assessing the efficacy with respect to clinical response rate of a combination of lurbinectedin and berzosertib as treatment of participants with recurrent SCLC and HGNEC.

Participants will receive lurbinectedin on day 1 and berzosertib on days 1 and 2, administered every 21 days (1 cycle), until disease progression or development of intolerable side effects.

Blood, hair follicles, and tumor will be collected at various time points to support the exploratory objectives.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Both Phase I and Phase II:
* >= 18 years of age.
* ECOG performance status <= 2
* Measurable disease, per RECIST 1.1. Individuals with evaluable, but not measurable disease will be eligible for Phase I.
* Adequate organ functions

  * Hemoglobin >= 9.0 g/dL
  * Absolute neutrophil count >= 1.5x10^9/L
  * Platelets >= 100x10^9/L
  * Total Bilirubin <= 2.0 mg/dL
  * Transaminases <= 2 x ULN or if liver metastases were present, <= 3 x ULN
  * Creatinine <= 1.5 mg/dL or creatinine clearance by Cockcroft-Gault formula >= 60 mL/min
* Ability to understand and the willingness to sign a written informed consent document.
* Individuals of child-bearing potential (IOCBP) and individuals able to father a child must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during study participation and for 6 months after the last dose of berzosertib/lurbinectedin for IOCBP and for 4 months after lurbinectedin or 3 months after berzosertib for individuals able to father children.

Phase I:

* Histologically confirmed advanced solid cancers will be eligible.
* At least one prior chemotherapy

Phase II:

- Histological confirmation of SCLC or HGNEC. Although NCI confirmation of pathology is not required prior to starting treatment, every effort will be made to obtain outside pathology to be reviewed by an NCI pathologist.

EXCLUSION CRITERIA:

* Individuals with tumor amenable to potentially curative therapy.
* Currently receiving any other investigational agents.
* Received chemotherapy, or undergone major surgery within the prior 2 weeks and radiotherapy within the last 24 hours.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to (study agent) or other agents used in study.
* Symptomatic brain metastases will be excluded from trial secondary to poor prognosis. However, individuals who have had treatment for their brain metastasis and whose brain disease is stable without steroid therapy for 1 week or on physiologic doses of steroids may be enrolled.
* Requirement for any medications or substances that are strong inhibitors or inducers of CYP3A during the course of the study are ineligible.
* Evidence of severe or uncontrolled systemic disease, or any concurrent condition, which could compromise participation in the study, including, but not limited to, active or uncontrolled infection, immune deficiencies, Hepatitis B, Hepatitis C, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, stroke/cerebrovascular accident within the past 6 months, or psychiatric illness/social situations which would jeopardize compliance with the protocol.
* HIV-positive on or off combination antiretroviral therapy are ineligible.
* Pregnant individuals are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
MTD | Phase I
  Maximum tolerated dose (MTD) of lurbinectedin in combination with berzosertib.
Clinical response rate | Phase II
  - Fraction of participants who experience a PR or CR in each cohort reported along with a 95% confidence interval. - Overall response rate for both cohorts combined, along with a 95% confidence interval.

SECONDARY OUTCOMES:
Safety and tolerability | Phase I
  Dose level Adverse Events (AE) per CTCAE v5.0, by type and grade of toxicity.
Pharmacodynamic markers of response | Phase I
  GammaH2ax and POLII as possible markers for pharmacodynamic activity and evaluation of changes in the markers between baseline and end of treatment vs. response
Pharmacokinetic profile of Berzosertib and Lurbinectedin | Phase I
  This will be evaluated using descriptive methods and reported as exploratory results. If any statistical tests are performed in these analyses, the results will be presented without adjustment for multiple comparisons but reported in the context of the number of tests performed.
Progression-free survival (PFS) | Phase II
  - Progression free survival will be determined from the on-study date until date of progression or death without progression, separately by cohort.
Overall survival (OS) | Phase II
  - Overall survival determined from the on-study date until date of death or last follow-up, separately by phase II cohort.
Duration of response | Phase II
  Duration of response to the combination in both platinum sensitive and refractory participants
Safety and tolerability of the MTD | Phase II
  Grades and types of toxicity will be reported for all patients treated at the DLT.

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Derived] Schultz CW, Zhang Y, Elmeskini R, Zimmermann A, Fu H, Murai Y, Wangsa D, Kumar S, Takahashi N, Atkinson D, Saha LK, Lee CF, Elenbaas B, Desai P, Sebastian R, Sharma AK, Abel M, Schroeder B, Krishnamurthy M, Kumar R, Roper N, Aladjem M, Zenke FT, Ohler ZW, Pommier Y, Thomas A. ATR inhibition augments the efficacy of lurbinectedin in small-cell lung cancer. EMBO Mol Med. 2023 Aug 7;15(8):e17313. doi: 10.15252/emmm.202217313. Epub 2023 Jul 25. PMID 37491889
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000176-C.html